CLINICAL TRIAL: NCT01436201
Title: Effect of Dulaglutide (LY2189265) on the Pharmacokinetics of Digoxin in Healthy Subjects
Brief Title: A Study of the Effect of Dulaglutide on How Body Handles Digoxin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11550; H9X-MC-GBCR (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Digoxin; dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Digoxin + Dulaglutide (Experimental): Digoxin: Two 0.5-milligram (mg) doses, oral, 12 hours apart on Day 1 (1 mg total on Day 1); 0.25 mg, oral, once daily on Day 2 to Day 17.
  Dulaglutide (LY2189265): 1.5 mg, subcutaneous injection, once on Day 8 and once on Day 15.
  Interventions: Drug: Digoxin; Biological: Dulaglutide

INTERVENTIONS:
Drug: Digoxin — Administered orally
Biological: Dulaglutide — Administered as subcutaneous injection
  Other Names: LY2189265

SUMMARY:
The purpose of this study is to study how the body processes digoxin and the effect of dulaglutide on how digoxin is processed by the body. Information about any side effects that may occur will also be collected.

This study is for research purposes only and is not intended to treat any medical condition. This research study requires that a blood sample be obtained and stored for future research involving genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Male participants with female partners of child-bearing potential, or partners who are pregnant or breastfeeding, agree to use a reliable method of contraception from the time of the first dose until 3 months after the last dose of investigational product, as determined by the investigator. The method may be one of the following:

  * Condom with spermicidal agent
  * Male participant sterilization
  * True abstinence (which is in line with the participant's usual lifestyle choice; withdrawal or calendar methods are not considered acceptable)
* Female participants not of child-bearing potential (that is, they are postmenopausal or permanently sterilized [such as, tubal occlusion, hysterectomy, bilateral salpingectomy]). Such participants will not be required to use contraception but must test negative for pregnancy at the time of enrolment. Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) or at least 1 year of spontaneous amenorrhea, with follicle stimulating hormone (FSH) ≥40 milli-international units per milliliter (mIU/mL)
* Female participants who have undergone sterilization by tubal ligation agree to use a condom in conjunction with spermicidal gel, foam, cream, film or suppository from the time of screening until 3 months after the last dose of investigational product. Such participants must also test negative for pregnancy at the time of enrolment
* Have a body mass index (BMI) of 18.5 to 32.0 kilogram per square meter (kg/m^2), inclusive, at screening
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator (potassium, magnesium, and calcium values must be within the normal range)
* Have normal renal function defined as an estimated creatinine clearance (CrCl) of ≥80 milliliter per minute (mL/min)
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study restrictions
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to glucagon like peptide-1 (GLP-1)-related compounds including dulaglutide (LY2189265) or to digoxin, related compounds or any components of either formulation
* Are participants who have previously completed or withdrawn from this study or any other study investigating dulaglutide in the 3 months prior to screening or have received glucagon-like peptides or incretin mimetics in the 3 months prior to screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) (such as, first, second, or third degree atrioventricular [AV] block, prolonged corrected QT [QTc] interval, sinus tachycardia, sinus bradycardia, atrial fibrillation, or sinus node disease) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history of significant dysrhythmias or AV block
* Have an abnormal blood pressure (after at least 5 minutes sitting) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of cardiac, respiratory, hepatic, renal, endocrine (such as, hypothyroidism), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or gastrointestinal disorder, for example relevant esophageal reflux or gall bladder disease, or any gastrointestinal disease which impacts gastric emptying (GE) (such as, gastric bypass surgery, pyloric stenosis, with the exception of appendectomy) or could be aggravated by GLP-1 analogs. Participants with dyslipidemia, and participants who had cholecystolithiasis (removal of gall stones) and/or cholecystectomy (removal of gall bladder) in the past, with no further sequelae, may be included in the study at the discretion of the screening physician
* Show evidence of significant active neuropsychiatric disease
* Have family history of medullary thyroid cancer (MTC) or a genetic condition that predisposes to MTC
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Have used or intend to use over-the-counter medication other than acetaminophen within 7 days prior to dosing or prescription medication (with the exception of vitamin/mineral supplements) within 14 days prior to dosing, or have used St John's Wort within 14 days prior to dosing
* Have donated blood of more than 500 mL within the month prior to screening
* Have an average weekly alcohol intake that exceeds 21 units per week (males) 14 units per week (females), or are unwilling to stop alcohol consumption from screening through follow-up (1 unit = 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Are smokers
* Have a history of cancer with the past 20 years, with the exception of basal cell or squamous cell skin cancer, or treated cervical carcinoma in situ
* Intend to consume grapefruit within 7 days prior to dosing
* Are participants who, in the opinion of the investigator, are in any way unsuitable to participate in the study
* Have any medical conditions, medical history or are taking any medication which are contraindicated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

REFERENCES:
- [Derived] de la Pena A, Cui X, Geiser J, Loghin C. No Dose Adjustment is Recommended for Digoxin, Warfarin, Atorvastatin or a Combination Oral Contraceptive When Coadministered with Dulaglutide. Clin Pharmacokinet. 2017 Nov;56(11):1415-1427. doi: 10.1007/s40262-017-0531-7. PMID 28357715

RESULTS

PARTICIPANT FLOW:
Groups:
- Digoxin + Dulaglutide: Digoxin: Two 0.5-milligram (mg) doses, administered orally, 12 hours apart on Day 1 (1 mg total on Day 1); 0.25 mg, orally, once daily on Day 2 to Day 17.
  Dulaglutide (LY2189265): 1.5 mg, subcutaneous injection, once on Day 8 and once on Day 15.
Period: Overall Study
Arm/Group | Digoxin + Dulaglutide
Started | 24
Received at Least 1 Dose of Study Drug | 24
Completed | 20
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Digoxin + Dulaglutide
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of Digoxin
Time Frame: Predose (Digoxin) and up to 24 hours postdose on Days 7, 10, and 17
Population: Participants who received at least one dose of study drug (digoxin or dulaglutide) with evaluable digoxin AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms times hours/milliliter
Groups:
- Digoxin Only: Digoxin: Two 0.5-milligram (mg) doses, administered orally, 12 hours apart on Day 1 (1 mg total on Day 1); 0.25 mg, orally, once daily on Day 2 to Day 7.
- Digoxin + Dulaglutide: Digoxin: Two 0.5-milligram (mg) doses, administered orally, 12 hours apart on Day 1 (1 mg total on Day 1); 0.25 mg, orally, once daily on Day 8 to Day 17.
  Dulaglutide (LY2189265): 1.5 mg, subcutaneous injection, once on Day 8 and once on Day 15.
Arm/Group | Digoxin Only | Digoxin + Dulaglutide
Number analyzed (Participants) | 21 | 21
nanograms times hours/milliliter
  Day 7 | 16.8 (25) | NA (NA) — Participants had not received dulaglutide dose at Day 7.
  Day 10 | NA (NA) — Participants received digoxin + dulaglutide dose at Day 10 (not digoxin only). | 16.1 (26)
  Day 17 (n=20) | NA (NA) — Participants received digoxin + dulaglutide dose at Day 17 (not digoxin only). | 16.3 (32)

2. Primary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of Digoxin
Time Frame: Predose (Digoxin) and up to 24 hours postdose on Days 7, 10, and 17
Population: Participants who received at least one dose of study drug (digoxin or dulaglutide) with evaluable digoxin Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | Digoxin Only | Digoxin + Dulaglutide
Number analyzed (Participants) | 21 | 21
nanograms per milliliter
  Day 7 | 1.71 (27) | NA (NA) — Participants had not received dulaglutide dose at Day 7.
  Day 10 | NA (NA) — Participants received digoxin + dulaglutide dose at Day 10 (not digoxin only). | 1.34 (40)
  Day 17 (n=20) | NA (NA) — Participants received digoxin + dulaglutide dose at Day 17 (not digoxin only). | 1.42 (42)

3. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Drug Concentration (Tmax) of Digoxin
Time Frame: Predose (Digoxin) and up to 24 hours postdose on Days 7, 10, and 17
Population: Participants who received at least one dose of study drug (digoxin or dulaglutide) with evaluable digoxin Tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | Digoxin Only | Digoxin + Dulaglutide
Number analyzed (Participants) | 21 | 21
hours
  Day 7 | 1.00 [0.50 to 1.50] | NA [NA to NA] — Participants had not received dulaglutide dose at Day 7.
  Day 10 | NA [NA to NA] — Participants received digoxin + dulaglutide dose at Day 10 (not digoxin only). | 1.50 [1.00 to 6.00]
  Day 17 (n=20) | NA [NA to NA] — Participants received digoxin + dulaglutide dose at Day 17 (not digoxin only). | 1.50 [1.00 to 4.00]

ADVERSE EVENTS:
Groups:
- Digoxin: Digoxin: Two 0.5-milligram (mg) doses, administered orally, 12 hours apart on Day 1 (1 mg total on Day 1); 0.25 mg, orally, once daily on Day 2 to Day 7.
Arm/Group | Digoxin | Digoxin + Dulaglutide
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 13/24 | 16/21
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin (N=24) | Digoxin + Dulaglutide (N=21)
Atrioventricular block first degree (Cardiac disorders) | 4 (5) | 6 (6)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 7 (9)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (2)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Vessel puncture site reaction (General disorders) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 6 (11)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days